CLINICAL TRIAL: NCT06503458
Title: Sickle Cell Disease Patient Reported Outcomes in Adult Participants Aged ≥18 Years of Age On and Off Hydroxyurea
Brief Title: A Low-Interventional Study of an Electronic Sickle Cell Disease Patient Reported Outcomes in Sickle Cell Participants
Status: Terminated | Type: Observational
Why Stopped: Low enrollment, cohorts were not able to be filled
Sponsor: Sanguine Biosciences (Industry)
Collaborators: Pfizer (Industry)
Responsible Party: Sponsor
Other Study IDs: C4071008
Record Dates: First submitted 2022-02-08; First posted 2024-07-16 (Actual); Last update posted 2024-07-16 (Actual); Status verified 2024-07

CONDITIONS: Sickle Cell Disease; Sickle Cell Anemia
Keywords: Sickle Cell Disease; Sickle Cell Anemia; SCD
MeSH Terms: conditions — Anemia, Sickle Cell

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Control Group: 1. Have experienced ≥1 episode(s) of MU VOC requiring documented unplanned medical intervention (eg, clinic, physician's office, emergency room or admission) requiring opioid or IV non-steroidal anti-inflammatory drug treatment within 12 months prior to Screening.
  2. Participant has no history of past treatment with HU unless the reason for discontinuation was pregnancy (or pregnancy of a partner).
  3. Data available for number of MU VOC(s) during the 12-month interval prior to Screening and a value for %HbF collected subsequent to 1 year of age in the absence of recent transfusion27(see Inclusion Criteria #2 - All Groups)
- HU Treatment Group: 1. Have experienced ≥1 episode(s) of MU VOC requiring documented unplanned medical intervention (eg, clinic, physician's office, emergency room or admission) requiring opioid or IV non-steroidal anti-inflammatory drug treatment within12 months prior to initiation of HU.
  2. Must be on a stable dose of HU ≥8 weeks prior to Day 1 with the intent of remaining on the same dose throughout the study, unless adjustments are medically necessary due to bone marrow suppression, in accordance with published guidelines.
  3. Data available for number of MU VOC(s) during the 12-month interval prior to initiation of HU treatment and a value for %HbF collected subsequent to 1 year of age, prior to initiation of HU treatment and in the absence of recent transfusion27(see Inclusion Criteria #2 - All Groups).

SUMMARY:
The purpose of this study is to learn more about painful crisis in people with Sickle Cell Disease. For this reason, Pfizer is conducting a study to understand how people with Sickle Cell Disease feel on a daily basis, treat these painful episodes including if they treat themselves at home or go to a doctor's office/emergency room, as well as the types of medications that are taken during these episodes.

DETAILED DESCRIPTION:
Pfizer is developing an ePRO that is completed on a daily basis using a diary to comprehensively self-report VOCs in participants with SCD and its impact on their lives.This is a prospective, low-intervention study to evaluate the responsiveness of the SCD ePRO in a therapeutic setting. Efficacy of drugs intended to reduce the frequency of VOC has historically been assessed based on frequency of VOC with an operational definition for VOC that requires MU, an endpoint approach that is limited in its utility for assessing benefit of therapeutic interventions across the totality of the disease experience. Thus, despite current available treatments, many patients with SCD still experience VOCs and there remains a significant unmet medical need and an opportunity to improve on existing endpoints. While previous studies have been conducted to consider this endpoint, they have not been conducted in a therapeutic setting and therefore unable to assess the responsiveness of theSCD ePRO.1,2This study aims to assess the responsiveness of the patient-reported endpoints in participants with SCD who are not on a disease modifying therapy versus those who are on the disease modifying treatment HU.

ELIGIBILITY:
Inclusion Criteria - Control Group

1. Have experienced ≥1 episode(s) of MU VOC requiring documented unplanned medical intervention (eg, clinic, physician's office, emergency room or admission) requiring opioid or IV non-steroidal anti-inflammatory drug treatment within 12 months prior to Screening.
2. Participant has no history of past treatment with HU unless the reason for discontinuation was pregnancy (or pregnancy of a partner).
3. Data available for number of MU VOC(s) during the 12-month interval prior to Screening and a value for %HbF collected subsequent to 1 year of age in the absence of recent transfusion.

Inclusion Criteria - HU Treatment Group

1. Have experienced ≥1 episode(s) of MU VOC requiring documented unplanned medical intervention (eg, clinic, physician's office, emergency room or admission) requiring opioid or IV non-steroidal anti-inflammatory drug treatment within12 months prior to initiation of HU.
2. Must be on a stable dose of HU ≥8 weeks prior to Day 1 with the intent of remaining on the same dose throughout the study, unless adjustments are medically necessary due to bone marrow suppression, in accordance with published guidelines.
3. Data available for number of MU VOC(s) during the 12-month interval prior to initiation of HU treatment and a value for %HbF collected subsequent to 1 year of age, prior to initiation of HU treatment and in the absence of recent transfusion.

Exclusion Criteria:

Medical Conditions:

1. Evidence or history of clinically significant hematological (non-SCD), renal, endocrine, pulmonary, gastrointestinal, cardiovascular (including overt stroke but excluding silent cerebral infarct), hepatic (excluding cholelithiasis), psychiatric or neurological disease as assessed from medical records.
2. Participants with any of the following acute or chronic infections or infection history as self-reported and/or assessed from medical records:

   * Fever ≤7 days of Screening;
   * Any infection requiring treatment with anti-infective drug(s) ≤2 weeks ofScreening;
   * COVID-19 infection unless 10 days have elapsed since symptoms first appeared, participant is without symptoms for ≥24 hours and is not experiencing post-COVID-19 symptoms.
3. Marked bone marrow suppression as evidenced by any of the following as per medical record: severe anemia, neutropenia (ANC <1500 mm3WBC), thrombocytopenia (platelet count <100,000 mm3) ≤8 weeks of Day 1.
4. Major surgery <3 months prior to Day 1 as self-reported and/or assessed from medical records or planned significant medical procedures during the study.
5. Females who are pregnant or plan to become pregnant during the study.
6. Other medical or psychiatric condition including cognitive impairment that prevents accurate reporting of pain and/or assessment of SCD symptoms, recent (within the past year) or active suicidal ideation/behavior, or laboratory abnormality that may increase the risk of study participation or, in the investigator's judgment, make the participant inappropriate for the study.

   Prior/Concomitant Therapy:
7. History of hematopoietic stem cell transplant or treatment with gene therapy as assessed from medical records.
8. History of simple transfusion ≤4 weeks of Day 1 as assessed from medical records.Prior/Concurrent Clinical Study Experience:
9. Previous administration with an investigational drug within 30days (or as determined by the local requirement) or 5half-lives preceding Day 1 (whichever is longer).

   Other Exclusions:
10. Active use of illicit drug as determined by the investigator.

    * A history or use of opioids will not be considered an exclusion if participant takes prescribed opioids for pain related to the underlying SCD.
    * A history or use of cannabinoids is not exclusionary.
11. History of alcohol abuse, dependence, or binge drinking within 6months of Screening as determined by the investigator.

    - Binge drinking is defined as a pattern of 5 (male)and 4 (female) or more alcoholic drinks in about 2 hours. As a general rule, alcohol intake should not exceed 14 units per week (1unit = 8 ounces (240 mL) beer, 1 ounce (30mL) of 40% spirit or 3 ounces (90 mL) of wine).
12. Unwilling or unable to comply with the criteria in the Lifestyle Considerations section (Section 5.3) of this protocol.
13. Investigator site staff or Pfizer employees directly involved in the conduct of the study, site staff otherwise supervised by the investigator, and their respective family members.

Lifestyle Considerations:

Investigational drugs are not permitted during the study.

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Study Population: Approximately 200 participants with SCD (HbS/S or HbS/β-thal) will be enrolled into two concurrentgroups, those who are either not on disease modifying treatment (control group[Group 1], approximately 150 participants) or on a stable dose of HU(HU treatment group[Group 2], approximately 50 participants), will be enrolled in this study.
Sampling Method: Non-Probability Sample
Enrollment: 52 (Actual)
Dates: Start 2022-01-19 (Actual); Primary Completion 2023-12-23 (Actual); Study Completion 2024-04-10 (Actual)

PRIMARY OUTCOMES:
Primary Objective #1: | 6 months
  To assess whether the effect of HU on frequency of physician-reported MU VOC is observed in the study population, the annualized rate reduction in those on HU as compared to matched participants in control group will be evaluated. The null hypothesis is that the annualized physician-reported MU VOC rate in HU treatment group is not different from one in control group.
Primary Objective #2 | 6 months
  To assess whether the effect of HU on frequency of patient-reported crisis rates (VOC Day rate and Patient-reported VOC Event rate) calculated using SCD ePRO is observed in the study population, the annualized rates reduction in HU treatment group as compared to matched participants in control group will be evaluated. The corresponding null hypotheses are that the annualized patient-reported crisis rates in HU treatment group are not different from ones in control group.

SECONDARY OUTCOMES:
Association Between Patient-Reported Crisis Rates and Physician-Reported MU VOC rate | 6 months
  Patient-reported crisis rates are determined by VOC Day rate and patient-reported VOC Event rate and is calculated using the SCD ePRO. These will be compared to physician-reported MU VOC rate to assess if there is an association between them. The assessment will be done in the matched sample, as well as in those in HU treatment group and in matched control group participants. The corresponding null hypotheses are that the annualized patient-reported crisis rates are not associated with physician-reported MU VOC.

CONTACTS AND LOCATIONS:
Locations (1):
- Sanguine Biosciences, Woburn, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No